CLINICAL TRIAL: NCT04247464
Title: Evaluation of Short-term Fasting Effects on Chemotherapy Toxicity and Efficacy
Brief Title: Short-term Fasting as an Enhancer of Chemotherapy: Pilot Clinical Study on Colorectal Carcinoma Patients
Acronym: CHEMOFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Collaborators: Hospital Infanta Sofia (Other); Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP PI-3536
Record Dates: First submitted 2020-01-14; First posted 2020-01-30 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Fasting
Keywords: Short-term Fasting; Colorectal Cancer; Chemotherapy; Toxicity; Immune response
MeSH Terms: conditions — Fasting; Intermittent Fasting; Colorectal Neoplasms | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard diet (No Intervention): The participants will follow an standard diet during the chemotherapy treatment
- Fasting (Experimental): The participants will follow a short-term fasting period for 44-48 hours, starting 24 hours before chemotherapy treatment
  Interventions: Procedure: Fasting

INTERVENTIONS:
Procedure: Fasting — Food intake restriction
  Arms: Fasting

SUMMARY:
This study will evaluate the ability of short-term fasting to reduce chemotherapy toxicity and enhance anti-tumour response in patients with colorectal carcinoma subjected to chemotherapy.

DETAILED DESCRIPTION:
Fasting for 24-48 hours during chemotherapy improves the response of the immune system against tumors and reduces chemotherapy toxicity through yet unknown mechanisms. The investigators have found that fasting induces the activation of p21, a protein that stops cell proliferation and plays important immune roles. The investigators hypothesize that p21 induction with short-term fasting enhances the immune anti-tumour response and reduces chemotherapy toxicity. To test this, half of the colorectal carcinoma (CRC) participants will follow 48 hours of fasting, 24 before and 24 after chemotherapy, under constant and specialized nutritional supervision. While the other half will follow a standard diet. A complete blood immunological profile at each chemotherapy cycle will be generated in collaboration with expert cytometrists, and gene expression, biochemical parameters, tumor evolution and toxicity markers will be measured. The investigators will (1) perform a complete analysis of immune cells to characterize the immune effects of fasting during chemotherapy; (2) analyze the effects of fasting on genes, metabolites and other molecules, to identify the responsible biological mechanisms, focusing on p21; (3) assess the reduction of chemotherapy toxicity in patients of colorectal carcinoma subjected to short-term fasting during chemotherapy.

Our project will further explore a safe, inexpensive, relatively unexplored and powerful nutritional intervention that can improve the quality of life and survival rates of millions of cancer patients: short-term fasting. Also, our project will have an important scientific impact, since previous reports have not yet described a clear mechanism explaining the beneficial effects of short-term fasting with chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Participants with malignant colorectal neoplasia
* Good metabolic state (BMI>22)
* Good nutritional tests
* Normal Haematological and biochemical parameters
* Normal renal and hepatic function
* No loss of weight during the chemotherapy treatment

Exclusion Criteria:

* BMI<22
* Pregnancy or lactating women
* Bad nutritional state
* 3% weigh loss during the last month or more than 5% in the last three months
* Diagnosis of type 2 diabetes mellitus or hypertension
* Diagnosed hepatic, renal or cardiovascular disease
* Respiratory of psychiatric disease
* Nausea or vomiting, gastrointestinal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in the Common Terminology Criteria for Adverse Events CTCAE 5.0 toxicity table score. | Baseline and after three weeks
  To evaluate changes in chemotherapy toxicity, the Common Terminology Criteria for Adverse Events (CTCAE) 5.0 toxicity table score will be calculated, taking into account different analysis and questionnaires on toxicity symptoms.
  Analysis will include:
  * Hematological analysis (erythrocytes, thrombocytes, white blood cells, Neutrophil/lymphocyte ratio and Platelet/lymphocyte ratio).
  * Biochemical analysis (sodium, potassium, calcium, phosphate, urea, creatinine, total protein, albumin, bilirubin, alkaline phosphatase, lactate dehydrogenase, alanine transaminase, aspartate transaminases, creatine kinase, troponin T, C Reactive Protein (CRP), cortisol and prealbumin)
  * Subjective symptoms obtained from health questionnaires (hunger, nausea, dizzying, weakness, diarrhea, constipation, gastroesophageal reflux disease)
Changes in the immune response | Baseline and after three weeks
  To evaluate the effect of short-term fasting on the immune response a complete immune phenotyping by flow cytometry will be done: cluster of differentiation 3 (CD3), cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8) (for T cells); cluster of differentiation 19 (CD19) (for B-cells), the high affinity Interleukin-2 receptor alpha subunit (CD45RA), CD62L (for T cell subsets: Memory, Effector); cluster of differentiation 25 (CD25) and cluster of differentiation 127 (CD127) (both for Treg cells); cluster of differentiation 11b C(D11b) (for granulocytes and macrophages); cluster of differentiation 14 (CD14) (for monocytes); cluster of differentiation antigen 16 (CD16), cluster of differentiation 56 (CD56) (NK cells); cluster of differentiation 15 (CD15) (for granulocytes and monocytes) markers will be analyzed
Changes in the correlation between chemotherapy response and p21 and/or other fasting genes expression in peripheral blood mononuclear cells (PBMCs) | Baseline and after three weeks
  The expression levels of p21 and/or fasting genes in peripheral blood mononuclear cells (PBMCs) will be correlated with toxicity parameters previously described in the primary outcome measure 1

SECONDARY OUTCOMES:
Subjective evaluation of tolerance to fasting | 48 hours of fasting, including 24 hours prior and 24 hours after chemotherapy administration.
  To evaluate the tolerance to fasting, participants will fill in a fasting tolerance test based on the symptoms they feel, this will result in a final score of tolerance to fasting.
Changes in glycemia in response to fasting | Baseline and after three weeks
  Glucose levels (milligrams per milliliter) will be measured with a kit from Abbott Laboratories, by enzymatic spectrophotometric assays using an Architect instrument from Abbot Laboratories.
Changes in Free Fatty Acids levels in response to fasting | Baseline and after three weeks
  Free fatty acids levels (moles per milliliter) will be evaluated with a kit from Abbott Laboratories, by enzymatic spectrophotometric assays using an Architect instrument from Abbott Laboratories.
Changes in Insulin levels in response to fasting | Baseline and after three weeks
  Insulin levels (International Units per milliliter) will be measured with a kit from Abbott Laboratories, by luminescent immunoassay using the Architect instrument from Abbott Laboratories.
Changes ketone bodies in response to fasting | Baseline and after three weeks
  Ketone bodies concentration (moles per milliliter) will be measured with a kit from Sigma-Aldrich, by an enzymatic spectrophotometric assay using an microplate reader from Thermo Fisher.
Changes in gene expression in PBMCs after fasting | Baseline and after three weeks
  To evaluate changes in gene expression in PBMCs the following fasting genes will be analyzed by qRTPCR:
  * p21
  * Pyruvate Dehydrogenase Kinase 4 (PDK4)
  * Carnitine palmitoyltransferase 1 (CPT1)
  * Adipophilin (ADFP)
  * Solute carrier family 25, member 50 (SLC25A50)
Antitumoral response associated to fasting after chemotherapy treatment | Baseline and after three weeks
  To evaluate the clinical antitumoral response, different tumoral markers such as carcinoembryonic antigen (CEA) and Carbohydrate antigen (Ca 19.9) will be analyzed in serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Casado, MD, Principal Investigator — Hospital Universitario Infanta Sofia; Francisco Zambrana, MD, Principal Investigator — Hospital Universitario Infanta Sofia; Pablo J Fernandez-Marcos, PhD, Principal Investigator — IMDEA Food; Jaime Feliu, MD, Principal Investigator — Hospital Universitario La Paz; Nuria Rodríguez-Salas, MD, Principal Investigator — Hospital Universitario La Paz; Ismael Ghanem- Cañete, MD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- IMDEA Food, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mattson MP, Longo VD, Harvie M. Impact of intermittent fasting on health and disease processes. Ageing Res Rev. 2017 Oct;39:46-58. doi: 10.1016/j.arr.2016.10.005. Epub 2016 Oct 31. PMID 27810402
- [Background] Duan W, Guo Z, Jiang H, Ware M, Mattson MP. Reversal of behavioral and metabolic abnormalities, and insulin resistance syndrome, by dietary restriction in mice deficient in brain-derived neurotrophic factor. Endocrinology. 2003 Jun;144(6):2446-53. doi: 10.1210/en.2002-0113. PMID 12746306
- [Background] Arumugam TV, Phillips TM, Cheng A, Morrell CH, Mattson MP, Wan R. Age and energy intake interact to modify cell stress pathways and stroke outcome. Ann Neurol. 2010 Jan;67(1):41-52. doi: 10.1002/ana.21798. PMID 20186857
- [Background] Arnason TG, Bowen MW, Mansell KD. Effects of intermittent fasting on health markers in those with type 2 diabetes: A pilot study. World J Diabetes. 2017 Apr 15;8(4):154-164. doi: 10.4239/wjd.v8.i4.154. PMID 28465792
- [Background] Safdie FM, Dorff T, Quinn D, Fontana L, Wei M, Lee C, Cohen P, Longo VD. Fasting and cancer treatment in humans: A case series report. Aging (Albany NY). 2009 Dec 31;1(12):988-1007. doi: 10.18632/aging.100114. PMID 20157582
- [Background] Raffaghello L, Lee C, Safdie FM, Wei M, Madia F, Bianchi G, Longo VD. Starvation-dependent differential stress resistance protects normal but not cancer cells against high-dose chemotherapy. Proc Natl Acad Sci U S A. 2008 Jun 17;105(24):8215-20. doi: 10.1073/pnas.0708100105. Epub 2008 Mar 31. PMID 18378900
- [Background] Tinkum KL, Stemler KM, White LS, Loza AJ, Jeter-Jones S, Michalski BM, Kuzmicki C, Pless R, Stappenbeck TS, Piwnica-Worms D, Piwnica-Worms H. Fasting protects mice from lethal DNA damage by promoting small intestinal epithelial stem cell survival. Proc Natl Acad Sci U S A. 2015 Dec 22;112(51):E7148-54. doi: 10.1073/pnas.1509249112. Epub 2015 Dec 7. PMID 26644583
- [Background] Di Biase S, Lee C, Brandhorst S, Manes B, Buono R, Cheng CW, Cacciottolo M, Martin-Montalvo A, de Cabo R, Wei M, Morgan TE, Longo VD. Fasting-Mimicking Diet Reduces HO-1 to Promote T Cell-Mediated Tumor Cytotoxicity. Cancer Cell. 2016 Jul 11;30(1):136-146. doi: 10.1016/j.ccell.2016.06.005. PMID 27411588
- [Background] Pietrocola F, Pol J, Vacchelli E, Rao S, Enot DP, Baracco EE, Levesque S, Castoldi F, Jacquelot N, Yamazaki T, Senovilla L, Marino G, Aranda F, Durand S, Sica V, Chery A, Lachkar S, Sigl V, Bloy N, Buque A, Falzoni S, Ryffel B, Apetoh L, Di Virgilio F, Madeo F, Maiuri MC, Zitvogel L, Levine B, Penninger JM, Kroemer G. Caloric Restriction Mimetics Enhance Anticancer Immunosurveillance. Cancer Cell. 2016 Jul 11;30(1):147-160. doi: 10.1016/j.ccell.2016.05.016. PMID 27411589
- [Background] Lopez-Guadamillas E, Fernandez-Marcos PJ, Pantoja C, Munoz-Martin M, Martinez D, Gomez-Lopez G, Campos-Olivas R, Valverde AM, Serrano M. p21Cip1 plays a critical role in the physiological adaptation to fasting through activation of PPARalpha. Sci Rep. 2016 Oct 10;6:34542. doi: 10.1038/srep34542. PMID 27721423
- [Background] Caffa I, D'Agostino V, Damonte P, Soncini D, Cea M, Monacelli F, Odetti P, Ballestrero A, Provenzani A, Longo VD, Nencioni A. Fasting potentiates the anticancer activity of tyrosine kinase inhibitors by strengthening MAPK signaling inhibition. Oncotarget. 2015 May 20;6(14):11820-32. doi: 10.18632/oncotarget.3689. PMID 25909220
- [Background] Bouwens M, Afman LA, Muller M. Fasting induces changes in peripheral blood mononuclear cell gene expression profiles related to increases in fatty acid beta-oxidation: functional role of peroxisome proliferator activated receptor alpha in human peripheral blood mononuclear cells. Am J Clin Nutr. 2007 Nov;86(5):1515-23. doi: 10.1093/ajcn/86.5.1515. PMID 17991667